CLINICAL TRIAL: NCT01274468
Title: Tumor Markers in Lung Cancer
Status: Completed | Type: Observational
Sponsor: University of Oklahoma (Other)
Responsible Party: Principal Investigator, Gary Kinasewitz, Principal Investigator, University of Oklahoma
Other Study IDs: 14781
Record Dates: First submitted 2010-05-20; First posted 2011-01-11 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2012-08

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Lung biopsy
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to determine if DCAMLK1 can be measured in the endobronchial biopsy specimens and bronchial washings from patients with lung cancer.

DETAILED DESCRIPTION:
DCAMLK1 is a Ca2+ - ca/modulin (CaM) - dependent protein kinase that is a marker of stem cells in colonic crypts. Mutations within the stem cell population are thought to be responsible for the development of most colorectal carcinomas and studies have shown that DCAMLK1 is highly expressed in these tumors. Since the lung is an embryological development of the foregut, we speculate that DCAMLK1 will also be upregulated in lung cancers. The aim of this pilot study is to determine if DCAMLK1 can be measured in the endobronchial biopsy specimens and bronchial washings from patients with lung cancer.

This is a prospective study in 10 patients with lung masses suspected to be malignant who are scheduled for diagnostic bronchoscopy.

Patients with lung masses scheduled for diagnostic bronchoscopy will be included if they can give informed consent to participate and the diagnostic portion of the bronchoscopy has been uncomplicated. Patients considered to be at high risk during bronchoscopy because of either abnormal blood gases (Pco2 > 50 mmHg or PaO2 < 70 mmHg on oxygen) or coagulopathy (platelets <100,000 or INR > 1.5) will be excluded.

If the preliminary results indicate this is feasible, we will then propose a larger study to examine DCAMLK1 distribution in normal and cancerous tissue as well as the predictive value of this biomarker.

ELIGIBILITY:
Inclusion Criteria:

* abnormality on chest x-ray that requires diagnosis and physically capable of undergoing bronchoscopy

Exclusion Criteria:

* <45 years
* Patients with severe abnormalities in blood gases and/or a coagulopathy will be excluded.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ten patients with an expected age >45 years
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2009-08; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Identification of DCAMLK1 in BAL and lung biopsy specimens. | After collection and analysis of specimens.

CONTACTS AND LOCATIONS:
Overall Officials: Gary T Kinasewitz, MD, Principal Investigator — OU Health Sciences Center
Locations (1):
- Veterans Affairs Medical Center, Oklahoma City, Oklahoma, United States

REFERENCES:
- [Background] Humphries A, Wright NA. Colonic crypt organization and tumorigenesis. Nat Rev Cancer. 2008 Jun;8(6):415-24. doi: 10.1038/nrc2392. Epub 2008 May 15. PMID 18480839